CLINICAL TRIAL: NCT05444972
Title: A Multi-Country, Real-World Study to Explore Treatment Patterns, Effectiveness and Healthcare Resource Utilization for Patients Diagnosed With Myelofibrosis Through Chart Review
Brief Title: A Study to Explore Treatment Patterns, Treatment Outcomes, Healthcare Resource Utilization in Adult Participants With Myelofibrosis Through Chart Review
Acronym: METER
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H23-122
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Cancer
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Undergoing Chart Review: Participants treated for myelofibrosis undergoing chart review.

SUMMARY:
Myelofibrosis (MF) is a rare blood cancer, characterized by extensive fibrosis (scarring) of the bone marrow. It is one of a group of cancers known as myeloproliferative neoplasms (MPNs) in which bone marrow cells that produce blood cells develop and function abnormally. This study will evaluate treatment patterns, treatment outcomes, healthcare resource utilization in adult participants with Myelofibrosis.

Data from approximately 1000 participants will be collected. No participants will be enrolled in this study.

Participants' charts will be reviewed. No drug will be administered as a part of this study. The duration of the observation period is up to 156 weeks.

There is no additional burden for participants in this trial. All visits must be completed prior to data extraction and participants will be followed for up to 156 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Treated for myelofibrosis (MF) [primary myelofibrosis (PMF) and secondary myelofibrosis (SMF)].
* Must have initiated their first treatment on or after the first date when ruxolitinib was approved in their country of residence and no later than 31 December 2021.

Exclusion Criteria:

- Having received MF treatment in a clinical trial setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants patients diagnosed with myelofibrosis and treated on or after the first date when ruxolitinib was approved in their country of residence and no later than 31 December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Time from Diagnosis of Myelofibrosis (MF) to Initial Treatment | Up to Week 156
  Time from diagnosis of MF to initial treatment.
Duration of Initial Treatment | Up to Week 156
  Duration of initial treatment.
Duration of Second Treatment | Up to Week 156
  Duration of second treatment.
Duration of Subsequent Treatments | Up to Week 156
  Duration of subsequent treatments.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (66):
- United States (4):
  - UAB Comprehensive Cancer Center /ID# 252767, Birmingham, Alabama
  - Wellness Oncology & Hematology /ID# 255591, West Hills, California
  - Brigham & Women's Hospital /ID# 254312, Boston, Massachusetts
  - Gabrail Cancer Center Research /ID# 252768, Canton, Ohio
- Argentina (3):
  - Instituto FIDES /ID# 245526, La Plata, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 244373, Ciudad Autonoma Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - Fundaleu /Id# 244371, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
- Australia (4):
  - Townsville University Hospital /ID# 246585, Douglas, Queensland
  - Royal Adelaide Hospital /ID# 246583, Adelaide, South Australia
  - Fiona Stanley Hospital /ID# 246584, Murdoch, Western Australia
  - Royal Perth Hospital /ID# 246586, Perth, Western Australia
- Brazil (2):
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein /ID# 247394, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo /ID# 247392, São Paulo
- Canada (7):
  - St. Paul's Hospital /ID# 249719, Vancouver, British Columbia
  - Nova Scotia Health /ID# 248393, Halifax, Nova Scotia
  - Juravinski Cancer Centre /ID# 251334, Hamilton, Ontario
  - Princess Margaret Cancer Centre /ID# 249748, Toronto, Ontario
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 250449, Lévis, Quebec
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 250563, Montreal, Quebec
  - Jewish General Hospital /ID# 250674, Montreal, Quebec
- Colombia (5):
  - Organizacion Clinica Bonnadona -PREVENIR S.A.S. /ID# 244589, Baranquilla, Atlántico
  - Coorp Hosp Juan Ciudad Sede Hospital Universitario Mayor Mederi /ID# 246108, Bogota DC, Cundinamarca
  - Fundacion Santa Fe de Bogota /ID# 244588, Bogota, Cundinamarca
  - Clínica Imbanaco S.A.S /ID# 248465, Cali
  - Hospital Pablo Tobon Uribe /ID# 244525, Medellín
- Greece (8):
  - General Hospital of Athens Laiko /ID# 246159, Athens, Attica
  - University General Hospital Attikon /ID# 246167, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 246163, Heraklion, Crete
  - General University Hospital of Alexandroupolis /ID# 246161, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 246165, Athens
  - University General Hospital of Ioannina /ID# 246160, Ioannina
  - METAXA Cancer Hospital of Piraeus /ID# 246164, Piraeus
  - University General Hospital of Patras /ID# 246162, RION Patras Achaia
- Italy (10):
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant Anna /ID# 245149, Cona, Ferrara
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 245335, Rome, Lazio
  - Azienda Ospedaliera di Perugia /ID# 245415, Perugia, Umbria
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 245716, Bologna
  - ASST Spedali civili di Brescia /ID# 244910, Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 244909, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 245566, Novara
  - Azienda Ospedaliera Universitaria Paolo Giaccone /ID# 245075, Palermo
  - ASST Sette Laghi /ID# 245443, Varese
  - Ospedale Belcolle /ID# 245726, Viterbo
- Mexico (3):
  - Hospital de Especialidades CMN SigloXXI /ID# 244748, Mexico City, Mexico City
  - Centro Regiomontano de Estudios Clínicos ROMA S.C /ID# 244750, Monterrey, Nuevo León
  - Hospital General de Mexico /ID# 244749, Mexico City
- Poland (4):
  - Krzysztof Mądry Praktyka Lekarska /ID# 250485, Warsaw, Masovian Voivodeship
  - Specjalistyczna Praktyka Lekarska Witold Prejzner /ID# 250516, Gdansk, Pomeranian Voivodeship
  - Joanna Góra-Tybor Specjalistyczna Praktyka Lekarska /ID# 250495, Lodz
  - Specjalistyczna Praktyka Lekarska Grzegorz Helbig /ID# 250515, Orzesze
- Portugal (3):
  - Centro Hospitalar e Universitario de Coimbra, EPE /ID# 244687, Coimbra
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 248203, Lisbon
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 244400, Porto
- Romania (4):
  - MedLife - Policlinica de Diagnostic Rapid /ID# 244395, Brasov, Brașov County
  - Spitalul Clinic Colentina /ID# 245620, Bucharest
  - Institutul Clinic Fundeni /ID# 245939, Bucharest
  - Institutul Oncologic Prof Dr I Chiricuta /ID# 244393, Cluj-Napoca
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 250092, Kaohsiung City
  - National Taiwan University Hospital /ID# 250093, Taipei
- Turkey (Türkiye) (7):
  - Gulhane Askeri Tip Academy /ID# 244134, Ankara
  - Hacettepe University Medical Faculty /ID# 244131, Ankara
  - Dicle Universitesi Tip /ID# 244137, Diyarbakır
  - Trakya University Medical Facu /ID# 244132, Edirne, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi /ID# 244133, Istanbul
  - Ege University Medical Faculty /ID# 244130, Izmir
  - Inonu University Medical Faculty /ID# 244135, Malatya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gupta V, Tomuleasa C, Barranco Lampon GI, Hou HA, Helbig G, Vachhani P, Symeonidis A, Haznedaroglu I, Galvez K, Tatsch F, Chopra AS, Zhang M, Vizkelety T, Murray B, Ross DM. Real-world treatment patterns and health care resource use for patients with myelofibrosis: results from the METER study. Blood Adv. 2025 Mar 11;9(5):1105-1116. doi: 10.1182/bloodadvances.2024014625. PMID 39729499